CLINICAL TRIAL: NCT01354964
Title: Effect of Vitamin D Repletion on Insulin Resistance and Systemic Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Meredith Hawkins, Professor of Medicine (Endocrinology), Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-225; 5K23RR023335-02 (NIH)
Record Dates: First submitted 2011-05-12; First posted 2011-05-17 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Insulin Resistance
Keywords: Glucose Metabolism Disorders; Insulin Resistance; Endocrine System; Vitamin D
MeSH Terms: conditions — Insulin Resistance; Glucose Metabolism Disorders | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): Participants received weekly oral vitamin D drops using a weight-based calculated dosage for up to six months.
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): Participants received weekly oral placebo drops (similar in taste and appearance to vitamin D) for up to six months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D
  Other Names: Vitamin D3 (cholecalciferol)
  Arms: Vitamin D
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research is to study the effects of Vitamin D supplementation on the body's response to insulin (a hormone that controls blood sugar), on inflammation, and on specific cells and processes in fat tissue.

DETAILED DESCRIPTION:
Over the last several years, studies have shown that low vitamin D levels may increase risk of developing Type 2 Diabetes. The investigators will administer vitamin D3 (cholecalciferol) to non-diabetic, insulin resistant subjects with vitamin D deficiency (total vitamin D levels <20 ng/ml) to increase the level of vitamin D3. The investigators will study the effects of increased Vitamin D on insulin action, adipose tissue inflammation, and on certain cells and processes in fat tissue.

Investigators will study participants with a procedure called a "pancreatic clamp" study. During the clamp procedure, glucose (a sugar) and insulin (a hormone produced in the pancreas that regulates the amount of glucose in the blood) are infused with an intravenous catheter, and blood samples are collected periodically throughout the procedure to measure blood sugar levels and the levels of several hormones that are found in the body and are related to glucose metabolism. Adipose tissue inflammation will be measured using the following inflammatory markers: IL-6, PAI-1, TNF-alpha, and iNOS.

ELIGIBILITY:
Inclusion Criteria:

* Serum 25(OH)D<20ng/ml
* Insulin Resistant based on HOMA-IR score of >3
* Able and willing to provide informed consent
* BMI 20-35

Exclusion Criteria:

* HIV/AIDS
* History of any cancer
* Sarcoidosis
* Alcohol or substance abuse
* Cushing's syndrome
* Primary hyperparathyroidism
* Nephrolithiasis
* Pregnancy or breastfeeding
* Regular visits to a tanning salon
* Hypercalcemia or hypocalcemia
* Untreated or uncontrolled hypertension
* Any chronic illness requiring medication, other than arthritis, hypertension and hyperlipidemia

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-03-13 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2015-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith A Hawkins, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D: Participants received weekly oral vitamin D drops using a weight-based calculated dosage for up to 6 months.
  .
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 11 | 8
Completed | 7 | 7
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — IV access issues | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vitamin D: Participants received weekly oral vitamin D drops using a weight-based calculated dosage for up to six months.
  .
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (10.7) | 47.3 (11.5) | 44.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 2 | 3 | 5
  Black or African American | 7 | 5 | 12
  Asian | 0 | 0 | 0
  Hispanic or Latino | 2 | 0 | 2
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 8 | 19
Hepatic Insulin Sensitivity [Mean (Standard Deviation); unit: mg/kg/min] — We examine the endogenous glucose production (EGP) to assess hepatic insulin sensitivity at baseline.
  mg/kg/min | 1.28 (0.65) | 1.10 (0.64) | 1.20 (0.63)
Peripheral Glucose Uptake [Mean (Standard Deviation); unit: mg/kg/min] — We examine the rate of glucose uptake to determine peripheral insulin sensitivity using rate of disappearance (Rd) of glucose.
  mg/kg/min | 5.99 (1.18) | 6.71 (2.33) | 6.29 (1.74)
Evaluated expression of pro-inflammatory gene TNF-α in macrophages [Mean (Standard Deviation); unit: Ratio of mRNA copy numbers (TNF-α/5HKGs)] — Adipose tissue macrophages will be isolated from subcutaneous abdominal adipose tissue, and will be quantified by fluorescence activated cell sorting (FACS) analysis. TNF-α gene expression will be examined by real-time polymerase chain reaction (rt-PCR) and will provide a measure of macrophage activation. The mRNA copy number is then compared with a reference gene copy number (5 commonly used house keeping genes [HKGs]) as a ratio, which is a measure of relative gene expression. Population: TNFα was measured in 6 participants in placebo group.
  Ratio of mRNA copy numbers (TNF-α/5HKGs)
    number analyzed (Participants) | 11 | 6 | 17
    (all) | 0.05 (0.03) | 0.02 (0.02) | 0.04 (0.03)
Evaluated expression of pro-inflammatory gene IL-6 in macrophages [Mean (Standard Deviation); unit: Ratio of mRNA copy numbers (IL-6/5HKGs)] — Adipose tissue macrophages will be isolated from subcutaneous abdominal adipose tissue, and will be quantified by fluorescence activated cell sorting (FACS) analysis. IL-6 gene expression will be examined by real-time polymerase chain reaction (rt-PCR) and will provide a measure of macrophage activation. The mRNA copy number is then compared with a reference gene copy number (5 commonly used house keeping genes [HKGs]) as a ratio, which is a measure of relative gene expression. Population: IL-6 was measured in 6 participants in placebo group.
  Ratio of mRNA copy numbers (IL-6/5HKGs)
    number analyzed (Participants) | 11 | 6 | 17
    (all) | 0.06 (0.05) | 0.04 (0.05) | 0.05 (0.05)
Evaluated expression of pro-inflammatory gene iNOS in macrophages [Mean (Standard Deviation); unit: Ratio of mRNA copy numbers (iNOS/5HKGs)] — Adipose tissue macrophages will be isolated from subcutaneous abdominal adipose tissue, and will be quantified by fluorescence activated cell sorting (FACS) analysis. iNOS gene expression will be examined by real-time polymerase chain reaction (rt-PCR) and will provide a measure of macrophage activation. The mRNA copy number is then compared with a reference gene copy number (5 commonly used house keeping genes [HKGs]) as a ratio, which is a measure of relative gene expression. Population: iNOS was measured in 6 participants in placebo group.
  Ratio of mRNA copy numbers (iNOS/5HKGs)
    number analyzed (Participants) | 11 | 6 | 17
    (all) | 0.007 (0.008) | 0.006 (0.005) | 0.007 (0.007)
Evaluated expression of pro-inflammatory gene PAI-1 in macrophages [Mean (Standard Deviation); unit: Ratio of mRNA copy numbers (PAI-1/5HKGs)] — Adipose tissue macrophages will be isolated from subcutaneous abdominal adipose tissue, and will be quantified by fluorescence activated cell sorting (FACS) analysis. PAI-1 gene expression will be examined by real-time polymerase chain reaction (rt-PCR) and will provide a measure of macrophage activation. The mRNA copy number is then compared with a reference gene copy number (5 commonly used house keeping genes [HKGs]) as a ratio which is a measure of relative gene expression. Population: PAI-1 was measured in 6 participants in placebo group.
  Ratio of mRNA copy numbers (PAI-1/5HKGs)
    number analyzed (Participants) | 11 | 6 | 17
    (all) | 0.03 (0.03) | 0.04 (0.03) | 0.03 (0.03)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Hepatic Insulin Sensitivity
Description: Endogenous glucose production (EGP) was assessed at each study visit to evaluate hepatic insulin sensitivity. Percent change between the EGP at baseline and second visit (after treatment for up to 3 months with Vitamin D to reach a target level of ≥30 ng/ml), and baseline and third visits (after treatment for up to 6 months with Vitamin D in order to reach a target level of ≥50 ng/ml) will be calculated.
Time Frame: 2nd clamp visit (after up to 3 months) and 3rd clamp visit (after up to 6 months)
Population: Hepatic insulin sensitivity was measured in 7 (out of 11) participants in the Vitamin D group and in 7 (out of 8) participants in the placebo group at the 3rd study visit due to loss to follow up, withdrawal, or difficulties in obtaining IV access.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Vitamin D: Participants received weekly oral vitamin D drops using a weight-based calculated dosage to reach a target level of ≥30 ng/ml at second visit and a goal level of ≥50 ng/ml at third visit.
- Placebo: Participants received weekly oral placebo drops (similar in taste and appearance to vitamin D).
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 11 | 8
percent change
  Percent change between baseline and 2nd visit | -19.2 (11.6) | 5.8 (22.5)
  Percent change between baseline and 3rd visit: number analyzed (Participants) | 7 | 7
  Percent change between baseline and 3rd visit | -33.66 (7.5) | 113.7 (65.5)

2. Secondary Outcome: Percent Change in Peripheral Glucose Uptake
Description: The rate of glucose uptake to determine peripheral insulin sensitivity was measured using the rate of disappearance (Rd) of glucose at each study visit. Percent change between the Rd at baseline and second visit (after treatment with Vitamin D for up to 3 months to target level of ≥30 ng/ml), and baseline and third visits (after treatment with Vitamin D for up to 6 months to target level of ≥50 ng/ml) will be calculated.
Time Frame: 2nd clamp visit (up to 3 months) and 3rd clamp visit (up to 6 months)
Population: Hepatic insulin sensitivity was measured in 7 (out of 11) participants in the Vitamin D group and in 6 (out of 8) participants in the placebo group at the 3rd study visit due to loss to follow up, withdrawal, or difficulties in obtaining IV access.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 11 | 8
percent change
  Percent change between baseline and 2nd visit | 0.48 (8.1) | -2.54 (5.8)
  Percent change between baseline and 3rd visit: number analyzed (Participants) | 7 | 6
  Percent change between baseline and 3rd visit | -0.98 (7.2) | 1.75 (10.1)

3. Secondary Outcome: Evaluated Expression of Pro-inflammatory Gene TNF-α
Description: Adipose tissue macrophages will be isolated from subcutaneous abdominal adipose tissue, and will be quantified by fluorescence activated cell sorting (FACS) analysis. TNF-α gene expression will be examined by real-time (rt-PCR) and will provide a measure of macrophage activation at baseline, at 2nd study visit (after treatment with Vitamin D to a goal level of ≥30 ng/ml), and at 3rd study visit (goal Vitamin D level of ≥50 ng/ml). The mRNA copy number is then compared with a reference gene copy number (5 commonly used house keeping genes [HKGs]) as a ratio, which is a measure of relative gene expression.
Time Frame: 2nd clamp visit (up to 3 months) and 3rd clamp visit (up to 6 months)
Population: TNF-α expression was measured in 7 (out of 11) participants in the Vitamin D group and in 4 (out of 8) participants in the placebo group at the 3rd study visit due to loss to follow up, withdrawal, or difficulties in obtaining IV access. Additionally, 2 participants in placebo group did not provide fat biopsy samples for the study.
Measure: Mean (Standard Error); unit: Ratio of mRNA copy numbers (TNF-α/5HKGs)
Groups:
- Placebo: Participants in this group were assigned to receive weekly oral placebo drops (similar in taste and appearance to vitamin D) for three months.
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 11 | 6
Ratio of mRNA copy numbers (TNF-α/5HKGs)
  TNF-α (2nd study visit) | 0.023 (0.006) | 0.021 (0.007)
  TNF-α (3rd study visit): number analyzed (Participants) | 7 | 4
  TNF-α (3rd study visit) | 0.036 (0.009) | 0.008 (0.003)

4. Secondary Outcome: Evaluated Expression of Pro-inflammatory Gene IL-6
Description: Adipose tissue macrophages will be isolated from subcutaneous abdominal adipose tissue, and will be quantified by fluorescence activated cell sorting (FACS) analysis. IL-6 gene expression will be examined by real-time (rt-PCR) and will provide a measure of macrophage activation at baseline, at 2nd study visit (after treatment with Vitamin D to a goal level of ≥30 ng/ml), and at 3rd study visit (goal Vitamin D level of ≥50 ng/ml). The mRNA copy number is then compared with a reference gene copy number (5 commonly used house keeping genes [HKGs]) as a ratio, which is a measure of relative gene expression.
Time Frame: 2nd clamp visit (up to 3 months) and 3rd clamp visit (up to 6 months)
Population: IL-6 expression was measured in 7 (out of 11) participants in the Vitamin D group. For the placebo group, 6 of the 8 participants provided fat biopsy samples for the 2nd visit, and 4 participants provided for the 3rd visit due to loss to follow up, withdrawal, or difficulties in obtaining IV access.
Measure: Mean (Standard Error); unit: Ratio of mRNA copy numbers (IL-6/5HKGs)
Groups:
- Vitamin D: Participants in this group were assigned to receive weekly oral vitamin D drops using a weight-based calculated dosage for three months.
  .
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 11 | 6
Ratio of mRNA copy numbers (IL-6/5HKGs)
  IL-6 (2nd study visit) | 0.019 (0.006) | 0.047 (0.018)
  IL-6 (3rd study visit): number analyzed (Participants) | 7 | 4
  IL-6 (3rd study visit) | 0.022 (0.007) | 0.050 (0.029)

5. Secondary Outcome: Evaluated Expression of Pro-inflammatory Gene iNOS
Description: Adipose tissue macrophages will be isolated from subcutaneous abdominal adipose tissue, and will be quantified by fluorescence activated cell sorting (FACS) analysis. iNOS gene expression will be examined by real-time (rt-PCR) and will provide a measure of macrophage activation at baseline, at 2nd study visit (after treatment with Vitamin D to a goal level of ≥30 ng/ml), and at 3rd study visit (goal Vitamin D level of ≥50 ng/ml). The mRNA copy number is then compared with a reference gene copy number (5 commonly used house keeping genes [HKGs]) as a ratio, which is a measure of relative gene expression.
Time Frame: 2nd clamp visit (up to 3 months) and 3rd clamp visit (up to 6 months)
Population: iNOS expression was measured in 7 (out of 11) participants in the Vitamin D group. For the placebo group, 6 of the 8 participants provided fat biopsy samples for the 2nd visit, and 4 participants provided for the 3rd visit due to loss to follow up, withdrawal, or difficulties in obtaining IV access.
Measure: Mean (Standard Error); unit: Ratio of mRNA copy numbers (iNOS/5HKGs)
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 11 | 6
Ratio of mRNA copy numbers (iNOS/5HKGs)
  iNOS (2nd study visit) | 0.004 (0.002) | 0.008 (0.005)
  iNOS (3rd study visit): number analyzed (Participants) | 7 | 4
  iNOS (3rd study visit) | 0.003 (0.001) | 0.005 (0.002)

6. Secondary Outcome: Evaluated Expression of Pro-inflammatory Gene PAI-1
Description: Adipose tissue macrophages will be isolated from subcutaneous abdominal adipose tissue, and will be quantified by fluorescence activated cell sorting (FACS) analysis. PAI-1 gene expression will be examined by real-time (rt-PCR) and will provide a measure of macrophage activation at baseline, at 2nd study visit (after treatment with Vitamin D to a goal level of ≥30 ng/ml), and at 3rd study visit (goal Vitamin D level of ≥50 ng/ml). The mRNA copy number is then compared with a reference gene copy number (5 commonly used house keeping genes [HKGs]) as a ratio, which is a measure of relative gene expression.
Time Frame: 2nd clamp visit (up to 3 months) and 3rd clamp visit (up to 6 months)
Population: PAI-1 expression was measured in 7 (out of 11) participants in the Vitamin D group. For the placebo group, 6 of the 8 participants provided fat biopsy samples for the 2nd visit, and 4 participants provided for the 3rd visit due to loss to follow up, withdrawal, or difficulties in obtaining IV access.
Measure: Mean (Standard Error); unit: Ratio of mRNA copy numbers (PAI-1/5HKGs)
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 11 | 6
Ratio of mRNA copy numbers (PAI-1/5HKGs)
  PAI-1 (2nd study visit) | 0.020 (0.008) | 0.032 (0.012)
  PAI-1 (3rd study visit): number analyzed (Participants) | 7 | 4
  PAI-1 (3rd study visit) | 0.008 (0.005) | 0.019 (0.008)

ADVERSE EVENTS:
Time Frame: Time enrolled in study (approximately 6 months)
Groups:
- Vitamin D: Participants in this group were assigned to receive weekly oral vitamin D drops using a weight-based calculated dosage for six months.
  .
- Placebo: Participants in this group were assigned to receive weekly oral placebo drops (similar in taste and appearance to vitamin D) for six months.
Arm/Group | Vitamin D | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/8
Other Adverse Events (participants affected / at risk) | 1/11 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D (N=11) | Placebo (N=8)
benign paroxysmal vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D (N=11) | Placebo (N=8)
pre-syncopal episode (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes